CLINICAL TRIAL: NCT02942602
Title: Effect of Lipid Modifying Drugs on HDL Function in Patients With Hyperlipidemia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 4-2013-0281
Record Dates: First submitted 2016-10-17; First posted 2016-10-24 (Estimated); Last update posted 2018-07-18 (Actual); Status verified 2018-07

CONDITIONS: Hyperlipidemia
MeSH Terms: conditions — Hyperlipidemias | interventions — Atorvastatin; Cholestyramine Resin; Docosahexaenoic Acids; Ezetimibe

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Atorvastatin 20 mg (Experimental): lipid lowering treatment
  Interventions: Drug: Atorvastatin 20 mg
- Cholestyramine 8 g (Experimental): lipid lowering treatment
  Interventions: Drug: Cholestyramine 8 g
- Omega-3 (EPA+DHA) 2 g (Experimental): lipid lowering treatment
  Interventions: Drug: Omega-3 2g
- Atorvastatin 5 mg + Ezetimibe 10 mg (Experimental): lipid lowering treatment
  Interventions: Drug: Concurrent with Atorvastatin 5 mg + Ezetimibe 10 mg
- Life style modification for management of dyslipidemia (Active Comparator)
  Interventions: Behavioral: Lifestyle modification

INTERVENTIONS:
Drug: Atorvastatin 20 mg — The patients who meet the 2013 American College of Cardiology/American Heart Association criteria for receiving lipid-lowering therapy will be randomized into 5 groups.
  Arms: Atorvastatin 20 mg
Drug: Cholestyramine 8 g — The patients who meet the 2013 American College of Cardiology/American Heart Association criteria for receiving lipid-lowering therapy will be randomized into 5 groups.
  Arms: Cholestyramine 8 g
Drug: Omega-3 2g — The patients who meet the 2013 American College of Cardiology/American Heart Association criteria for receiving lipid-lowering therapy will be randomized into 5 groups.
  Arms: Omega-3 (EPA+DHA) 2 g
Drug: Concurrent with Atorvastatin 5 mg + Ezetimibe 10 mg — The patients who meet the 2013 American College of Cardiology/American Heart Association criteria for receiving lipid-lowering therapy will be randomized into 5 groups.
  Arms: Atorvastatin 5 mg + Ezetimibe 10 mg
Behavioral: Lifestyle modification — The patients who meet the 2013 American College of Cardiology/American Heart Association criteria for receiving lipid-lowering therapy will be randomized into 5 groups.
  Arms: Life style modification for management of dyslipidemia

SUMMARY:
1) to test HDL function comprehensively in healthy and diseased individuals; 2) to evaluate if this test correlates with cardiovascular risk, independent of traditional risk factors; 3) and to differentiate effects of lipid-modifying or antiatherosclerotic drugs on HDL function and composition

ELIGIBILITY:
Inclusion Criteria:

* The patients who meet the 2013 American College of Cardiology/American Heart Association criteria for receiving lipid-lowering therapy
* Aged over 20
* Consent form signed

Exclusion Criteria:

* pregnant or lactating women
* subjects with familial hypercholesterolemia
* uncontrolled hypertension or DM
* Thyroid dysfunction
* Active liver disease (transaminase or bilirubin > 1.5 x NL)
* Serum creatinine > 2 mg/dL
* Included in other clinical trials within 3 months
* using of other medication: fish oil, fibric acid derivatives, niacin, systemic corticosteroid, thiazolidinedione

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2014-04-03 (Actual); Primary Completion 2016-05-23 (Actual); Study Completion 2016-05-23 (Actual)

PRIMARY OUTCOMES:
Cholesterol efflux capacity (%) | Change of HDL functions from baseline to 8 weeks
  [3H-cholesterol (µCi) in medium containing HDL/(3H-cholesterol {µCi} in medium containing HDL+µCi of 3H-cholesterol {µCi} in cells)] x 100
Endothelial NO production (Arbitrary unit) | up to 8 weeks
  measured with nitrate assay kit and expressed as relative amount compared to control (no HDL treatment sample)
VCAM-1 expression (Arbitrary unit) | up to 8 weeks
  western blotting of VCAM-1 protein and expressed as relative amount compared to control (no HDL treatment sample)
ROS generation (Arbitrary unit) | up to 8 weeks
  fluorescence intensity measurement using dichlorodihydrofluorescein diacetate and expressed as relative amount compared to control (no HDL treatment sample)

SECONDARY OUTCOMES:
ApoA-I | Change of HDL associated proteins from each patient at baseline and at 8 weeks
  quantitation of intensity of western blot and expresses as relative amount to control (no HDL treatment sample)
ApoA-II | Change of HDL associated proteins from each patient at baseline and at 8 weeks
  quantitation of intensity of western blot and expresses as relative amount to control (no HDL treatment sample)
ApoC-I | Change of HDL associated proteins from each patient at baseline and at 8 weeks
  quantitation of intensity of western blot and expresses as relative amount to control (no HDL treatment sample)
ApoC-II | Change of HDL associated proteins from each patient at baseline and at 8 weeks
  quantitation of intensity of western blot and expresses as relative amount to control (no HDL treatment sample)
ApoC-III | Change of HDL associated proteins from each patient at baseline and at 8 weeks
  quantitation of intensity of western blot and expresses as relative amount to control (no HDL treatment sample)

CONTACTS AND LOCATIONS:
Locations (1):
- Division of Cardiology, Department of Internal Medicine,, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lee CJ, Choi S, Cheon DH, Kim KY, Cheon EJ, Ann SJ, Noh HM, Park S, Kang SM, Choi D, Lee JE, Lee SH. Effect of two lipid-lowering strategies on high-density lipoprotein function and some HDL-related proteins: a randomized clinical trial. Lipids Health Dis. 2017 Feb 28;16(1):49. doi: 10.1186/s12944-017-0433-6. PMID 28245873